CLINICAL TRIAL: NCT01130233
Title: Randomized Controlled Trial Comparing the Bladder and Sexual Functions of Patients Who Undergo Laparoscopic and Robotic Assisted Resection for Rectal Cancer
Brief Title: Randomized Trial on Robotic Assisted Resection for Rectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Professor Wai Lun LAW, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 09-132
Record Dates: First submitted 2010-05-24; First posted 2010-05-25 (Estimated); Last update posted 2010-05-25 (Estimated); Status verified 2010-05

CONDITIONS: Rectal Cancer; Adenocarcinoma
Keywords: rectal cancer
MeSH Terms: conditions — Rectal Neoplasms; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- robotic (Experimental): robotic assisted rectal resection
  Interventions: Procedure: robotic assisted rectal resection
- laparoscopic (Active Comparator): laparoscopic rectal resection
  Interventions: Procedure: laparoscopic rectal resection

INTERVENTIONS:
Procedure: robotic assisted rectal resection — robotic assisted rectal resection
  Arms: robotic
Procedure: laparoscopic rectal resection — laparoscopic rectal resection
  Arms: laparoscopic

SUMMARY:
Hypothesis: the bladder and sexual functions can be better preserved in patients with robotic assisted rectal surgery

This is a randomized trial comparing the bladder and sexual function of patients who undergo laparoscopic and robotic assisted rectal resection for rectal cancer.

DETAILED DESCRIPTION:
This is a randomized trial comparing the bladder and sexual function of patients who undergo laparoscopic and robotic assisted rectal resection for rectal cancer

The primary objective of this study is to compare the bladder and sexual functions of patients who undergo laparoscopic and robotic assisted resection for rectal cancer through a randomized controlled trial.

The secondary outcome measures include

1. The operative outcome in terms of the complication rate, hospital stay and reoperation of the two groups;
2. The quality of life of the patients and the cost of the two groups
3. The quality of the resected specimens
4. The local recurrence rates at two years after the surgery

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven new case of rectal cancer with the lower border within 15 cm from anal verge
2. Age >18 years
3. Informed consent obtained
4. American Society of Anesthesiologist class 1-3
5. No contraindication to laparoscopic surgery
6. Acceptable operating risk

Exclusion Criteria:

1. Locally advanced fixed tumor with the need for exenterative surgery
2. Severe cardiac or pulmonary comorbidity rendering pneumoperitoneum hazardous
3. Multiple previous operations with the anticipation of dense peritoneal adhesions
4. No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2009-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Bladder function | one year
  Urodynamic Questionnaire

SECONDARY OUTCOMES:
tumor status | One year
  recurrence and survival
Quality of life | one year
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Wai Lun Law, MBBS, MS, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong